CLINICAL TRIAL: NCT04935866
Title: Optimal Brain Oxygenation in Neurologic Intensive Care Unit : The NeurO2 Study
Acronym: NeurO2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Canadian Critical Care Trials Group (Other); Canadian Traumatic Brain Injury Research Consortium (Unknown)
Responsible Party: Principal Investigator, Dr Alexis Turgeon, Professor, CHU de Quebec-Universite Laval
Other Study IDs: MP-20-2021-5673
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Brain Injuries; Near-Infrared Spectroscopy; Intensive Care Neurological Disorder; Anemia
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Brain Injuries; Anemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Near-infrared spectroscopy (NIRS) — Non invasive brain oxygenation monitoring with Near-Infrared Spectroscopy (NIRS) technology. Patients enrolled in the NeurO2 study will have bilateral NIRS sensors applied to the forehead according to manufacturer recommendations. Data will be monitored continuously throughout the study intervention in the parent trials (HEMOTION and SAHaRA trials) in the neurocritical care unit. Data will be extracted from the device at the end of the study period.

SUMMARY:
The NeurO2 study is a multicenter observational study looking at NIRS monitoring in neurocrocritically ill patients during the acute phase of care following an acute brain injury. The study is nested within the HEMOTION Trial and the SAHaRA Trial

DETAILED DESCRIPTION:
The NeurO2 study is a multicenter prospective study nested within two large-scale pragmatic randomized open blinded endpoint (PROBE) trials in neurocritically ill patients, the HEMOTION and the SAHaRa trials. These two trials are designed to compare a restrictive and a liberal transfusion strategies in critically ill patients with traumatic brain injury or subarachnoid hemorrhage. The NeurO2 will report on prospectively gathered regional cerebral oxygenation data (rSO2) from enrolled patients randomized to either the liberal or restrictive RBC transfusion strategy of their parent trials. The primary outcome will be 6-month neurologic function based on the GOSe. The established infrastructure of the trials will be used, including part of the data collection instruments and the outcome assessment team.

The NeurO2 study will achieve three separate but interconnected primary objectives: i) Evaluate if the cerebral hypoxemic burden as measured by NIRS during NICU stay, is associated with functional neurologic outcome (Glasgow Outcome Scale extended - GOSe) at 6 months, ii) Determine if the cerebral hypoxemic burden is impacted by red blood cell transfusion, iii) Determine if the level of response in cerebral hypoxemic burden after RBC transfusion is associated with the 6-month functional neurologic outcome (GOSe)

The secondary objectives are to evaluate whether the cerebral hypoxemic burden measured by NIRS is associated with other clinically relevant outcomes including ICU, hospital and 6-month mortality and hospital, ICU length of stay and quality of life.

ELIGIBILITY:
Inclusion criteria:

* Enrolment in one of the parent trials (HEMOTION or SAHaRA trials)
* HEMOTION trial (acute moderate of severe blunt traumatic brain injury (Glasgow Coma Score18 [GCS] ≤ 12))
* SAHaRA trial (acute subarachnoid hemorrhage as confirmed by treating neurosurgeon or neuro-interventionist and supported by blood in subarachnoid space resulting from a ruptured aneurysm)
* Adult patients (age ≥18 years old)
* Patients suffering from anemia (Hb ≤100 g/L)

Exclusion criteria:

* Contraindications or known objections to blood transfusions
* Active bleeding with hemodynamic instability at the time of enrollment
* Decision to withdraw or withhold life-sustaining therapies made
* NIRS monitoring not reliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized with a traumatic brain injury or with aneurysmal subarachnoid hemorrhage already enrolled in the HEMOTION Trial or the SAHaRA Trial
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale extended | 6 months
  The GOSe is an ordinal scale on 8 points evaluating the neurological functional outcome in neurocritically ill patients where 1 represents death and 8 the best possible outcome.

SECONDARY OUTCOMES:
Mortality | 6 months
  Incidence of mortality
Hospital length of stay | through study completion, an average of 6 months
  Duration of hospital stay for the index hospitalisation
ICU length of stay | through study completion, an average of 6 months
  Duration of intensive care unit (ICU) stay for the index hospitalisation
EQ-5D-5L | 6 months
  EQ-5D-5L is a standardised measure of health-related quality of life developed by the EuroQol Group. The EQ-5D-5L includes a 5-dimension questionnaire and an overall health question using a visual analogue scale (VAS). The 5 dimensions of the EQ-5D-5L are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is evaluated based on 5 levels (from the worst (1) to the best (5)). The overall health evaluation is based on a 100 point VAS where 100 means the optimal health

CONTACTS AND LOCATIONS:
Overall Officials: Alexis F Turgeon, MD MSc FRCPC, Principal Investigator — CHU de Québec-Universite Laval Research Center, Universite Laval; Shane W English, MD MSc FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - CHU de Québec - Université Laval (Hôpital de l'Enfant-Jésus), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- See also: Canadian Traumatic Brain Injury Research Consortium — https://www.ctrc-ccrt.ca